CLINICAL TRIAL: NCT02900170
Title: Can Rivaroxaban Lead to Anticoagulation-Related Nephropathy?
Status: Completed | Type: Observational
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Basma Abdulhadi, Medical Resident, Albert Einstein Healthcare Network
Other Study IDs: 4831
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Acute Kidney Injury
Keywords: Rivaroxaban, Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anticoagulation-Related Nephropathy (ARN) is a side effect of treatment with blood thinners which leads to kidney dysfunction. A recent review suggests that kidney function should be assessed (by measuring serum creatinine) serially in the first few months of starting a blood thinner. ARN is diagnosed when there is a decline in kidney function after starting the blood thinner and other possible causes of this decline have been excluded. ARN has mainly been studied in relation to the common blood thinner - warfarin, where the prevalence is variable but can be as high as 37% (approximately 1 in 3) in the patients at highest risk. The risk factors that make this side effect more likely include the presence of pre-existing kidney disease, high blood pressure, older age and diabetes mellitus. Studies have shown that the occurence of ARN can lead to an accelerated progression of pre-existing kidney disease and a 65% increase in the risk of death (mortality).

The non-vitamin K oral anticoagulants (NOACs) are a new group of drugs which have been recently approved for use as blood thinners. They have a faster onset of action compared to warfarin and unlike warfarin, they do not need frequent monitoring. Rivaroxaban is the most commonly prescribed NOAC at Einstein Medical Center Philadelphia. There are some case reports that other NOACs (such as dabigatran and apixaban) can lead to ARN, however there is no study that has determined the true incidence of ARN in NOACs. Our study is designed to find out the incidence of ARN in patients who are started on rivaroxaban.

The investigators intend to serially monitor the kidney function of 40 high risk patients who are recently started on rivaroxaban over a six month period. This will enable us to discover how many patients actually develop ARN after starting a NOAC. The information the investigators will obtain from this study will enable patients and health care providers make better decisions about using blood thinners. If the investigators find that the incidence of ARN with rivaroxaban is less common than that previously reported with warfarin, it can potentially make more patients use the NOACs and hence save them from the morbidity and mortality associated with ARN. Our study is unique because this will be the first study focused on ARN in one of the new blood thinners. The information the investigators get from this study will be a very important foundation for future studies.

DETAILED DESCRIPTION:
Anticoagulation-related nephropathy (ARN) is an understudied renal complication of anticoagulant therapy that is characterized by acute kidney injury (AKI) defined as an increase in baseline serum creatinine ≥ 0.3 mg/dL, without any alternate etiology, in the setting of a supra-therapeutic International Normalized Ratio (INR) greater than 3.0 [1-7]. ARN has mainly been studied in relation to warfarin, it usually occurs in the first two months of starting anticoagulant therapy and retrospective studies have estimated the prevalence to range from 16% to 37% [4-6]. The strongest risk factor for ARN is pre-existing chronic kidney disease (CKD); other risk factors include older age, diabetes mellitus and hypertension [1,4]. Patients with ARN have an accelerated progression of CKD and a retrospective study of more than 15,000 patients on warfarin showed a 65% increase in mortality in patients with ARN [4,6].

The non-vitamin K oral anticoagulants (NOACs) are replacing warfarin in the clinical setting for long term anticoagulation because of the advantages of faster, reliable onset of action, and unlike warfarin, they do not require dose-response monitoring [8-10]. Rivaroxaban is the most commonly prescribed NOAC at Einstein Medical Center Philadelphia. A few animal models and case reports have shown that these NOACs (particularly dabigatran and apixaban) can lead to deterioration of kidney function, but there is limited epidemiologic data on ARN in NOACs and the incidence of ARN in NOACs is unknown [11-14]. A proposed guideline to diagnose ARN recommends that serum creatinine and urinalysis be checked monthly in the first few months of anticoagulation [1]. Clinical trials that compared warfarin to NOACs specifically studied stroke risk and bleeding outcomes and did not document the incidence of ARN because they did not make these regular creatinine and urinalysis measurements in the first few months of anticoagulation [15-20]. Our study intends to make these necessary measurements in a selected group of high risk patients started on rivaroxaban and hence determine the incidence of ARN in this group.

This study will be the first epidemiological study using a prospective design to measure the incidence of ARN in a population receiving NOACs. Given the high morbidity and mortality associated with ARN, the findings will enhance patient safety, enabling patients and health providers to make informed decisions with their patients regarding the choice of anticoagulants. It will also establish baseline data that will serve as foundation for future studies.

The specific aims of this study will be to -

1. Determine the incidence of ARN in high risk patients on rivaroxaban. Hypothesis - the incidence of ARN in rivaroxaban is less than the previously reported incidence of ARN in warfarin.
2. Describe demographic and urinalysis-associated predictors of ARN in patients on rivaroxaban.

SIGNIFICANCE

Anticoagulant-related nephropathy (ARN) is a relatively new and underdiagnosed complication of anticoagulant therapy with the potential to accelerate chronic kidney disease and lead to increased mortality [4,6]. Brodsky, et al, performed a retrospective study of more than 15,000 subjects and showed that the 5-year Kaplan-Meier survival rate was significantly lower in the ARN cohort compared to the patients without ARN with a 65% increased risk of mortality [4]. This dramatic increase in mortality that is attributable to an episode of ARN in a patient taking an anticoagulant is the reason why this study is very significant.

The clinical trials that compared the NOACs to warfarin did not specifically study ARN and did not repeat creatinine and urinalysis testing in the first two to three months of therapy to establish possible ARN diagnosis [15-20]. In most of these studies, only baseline creatinine and creatinine levels 6 to 12 months later were analyzed, hence it is possible that ARN was under-diagnosed as most cases of ARN are detected in the first eight weeks of therapy. Our study aims to accurately capture ARN cases by making these measurements monthly in the first three months of starting the anticoagulant.

This study is pivotal because it will for the first time, define the incidence of ARN in patients on rivaroxaban therapy. If the investigators find that ARN incidence in patients started on rivaroxaban is less than that seen with warfarin, this can help support evidence that this NOAC is safer for the kidneys compared to warfarin and this data can enable us make evidence based decisions regarding the continued use of the medication to help our patients. If on the other hand the investigators find that the medication leads to ARN, then the investigators will be contributing important post-marketing surveillance data that can also help us make safety decisions about the use of the medication in the future.

INNOVATION

Previous studies on ARN have utilized retrospective study designs which have many epidemiological pitfalls including the cause versus effect bias and the inability to ascertain relative risk [1]. Our study is unique because the investigators intend to utilize a prospective epidemiological design to study this renal complication, a first in the study of ARN. This is important because ARN is a diagnosis of exclusion and hence a prospective study is able to more accurately define cases of the condition compared to the assumptions that are made in retrospective studies where further work up cannot be done in retrospect.

This will be the first epidemiological study focused on ARN in a NOAC. Even though NOACs are new, they are becoming ubiquitous and a mainstay in clinical practice and not just an alternative to warfarin. For example, the recent CHEST guidelines recommend them as first line therapy in the treatment of venous thromboembolism [8]. Hence it will be important to clearly delineate their effects on the kidneys.

OBJECTIVES

In summary, this is a proposal for a prospective study to investigate the incidence of anti-coagulant nephropathy, a dreaded renal complication of anticoagulation. Our literature search has shown that there are no prospective studies of this condition in the new oral anticoagulants and clinical trials did not perform the necessary testing in the appropriately timed interval to diagnose ARN. The investigators chose to study rivaroxaban, the most commonly prescribed NOAC in our academic medical center and they anticipate that the result of this study will contribute safety data that will lead to better care of our patients and great cost savings by avoiding the morbidity and mortality associated with renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* GFR ≤ 60 ml/L based on creatinine clearance
* Participant has been initiated on long term anticoagulation with rivaroxaban for atrial fibrillation within four weeks of recruitment

Exclusion Criteria:

* History of blood dyscrasias or active bleeding,
* History of hematuria
* Patients on dialysis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study designed to determine the incidence of ARN in 40 adult patients recently initiated on rivaroxaban at Einstein Medical Center Philadelphia.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basma Abdulhadi, MD, Principal Investigator — Einstein Medical Center
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler DS, Giugliano RP, Rangaswami J. Anticoagulation-related nephropathy. J Thromb Haemost. 2016 Mar;14(3):461-7. doi: 10.1111/jth.13229. Epub 2016 Feb 15. PMID 26670286
- [Background] Brodsky SV, Satoskar A, Chen J, Nadasdy G, Eagen JW, Hamirani M, Hebert L, Calomeni E, Nadasdy T. Acute kidney injury during warfarin therapy associated with obstructive tubular red blood cell casts: a report of 9 cases. Am J Kidney Dis. 2009 Dec;54(6):1121-6. doi: 10.1053/j.ajkd.2009.04.024. Epub 2009 Jul 4. PMID 19577348
- [Background] Holbrook AM, Pereira JA, Labiris R, McDonald H, Douketis JD, Crowther M, Wells PS. Systematic overview of warfarin and its drug and food interactions. Arch Intern Med. 2005 May 23;165(10):1095-106. doi: 10.1001/archinte.165.10.1095. PMID 15911722
- [Background] Brodsky SV, Nadasdy T, Rovin BH, Satoskar AA, Nadasdy GM, Wu HM, Bhatt UY, Hebert LA. Warfarin-related nephropathy occurs in patients with and without chronic kidney disease and is associated with an increased mortality rate. Kidney Int. 2011 Jul;80(2):181-9. doi: 10.1038/ki.2011.44. Epub 2011 Mar 9. PMID 21389969
- [Background] An JN, Ahn SY, Yoon CH, Youn TJ, Han MK, Kim S, Chin HJ, Na KY, Chae DW. The occurrence of warfarin-related nephropathy and effects on renal and patient outcomes in korean patients. PLoS One. 2013;8(4):e57661. doi: 10.1371/journal.pone.0057661. Epub 2013 Apr 1. PMID 23560034
- [Background] Brodsky SV, Collins M, Park E, Rovin BH, Satoskar AA, Nadasdy G, Wu H, Bhatt U, Nadasdy T, Hebert LA. Warfarin therapy that results in an International Normalization Ratio above the therapeutic range is associated with accelerated progression of chronic kidney disease. Nephron Clin Pract. 2010;115(2):c142-6. doi: 10.1159/000312877. Epub 2010 Apr 22. PMID 20413993
- [Background] Limdi NA, Beasley TM, Baird MF, Goldstein JA, McGwin G, Arnett DK, Acton RT, Allon M. Kidney function influences warfarin responsiveness and hemorrhagic complications. J Am Soc Nephrol. 2009 Apr;20(4):912-21. doi: 10.1681/ASN.2008070802. Epub 2009 Feb 18. PMID 19225037
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Eikelboom JW, Weitz JI. New anticoagulants. Circulation. 2010 Apr 6;121(13):1523-32. doi: 10.1161/CIRCULATIONAHA.109.853119. No abstract available. PMID 20368532
- [Background] Augoustides JG. Breakthroughs in anticoagulation: advent of the oral direct factor Xa inhibitors. J Cardiothorac Vasc Anesth. 2012 Aug;26(4):740-5. doi: 10.1053/j.jvca.2012.03.029. Epub 2012 May 17. PMID 22608466
- [Background] Ryan M, Ware K, Qamri Z, Satoskar A, Wu H, Nadasdy G, Rovin B, Hebert L, Nadasdy T, Brodsky SV. Warfarin-related nephropathy is the tip of the iceberg: direct thrombin inhibitor dabigatran induces glomerular hemorrhage with acute kidney injury in rats. Nephrol Dial Transplant. 2014 Dec;29(12):2228-34. doi: 10.1093/ndt/gft380. Epub 2013 Sep 5. PMID 24009280
- [Background] Moeckel GW, Luciano RL, Brewster UC. Warfarin-related nephropathy in a patient with mild IgA nephropathy on dabigatran and aspirin. Clin Kidney J. 2013 Oct;6(5):507-9. doi: 10.1093/ckj/sft076. Epub 2013 Sep 10. PMID 26120444
- [Background] Ware KM, Vance JC, Muni N, Hebert LA, Satoskar AA, Nadasdy G, Ivanov I, Nadasdy T, Rovin BH, Brodsky SV. Oral warfarin and the thrombin inhibitor dabigatran increase blood pressure in rats: hidden danger of anticoagulants? Am J Hypertens. 2015 Feb;28(2):182-9. doi: 10.1093/ajh/hpu129. Epub 2014 Jul 13. PMID 25023204
- [Background] Stollberger C, Finsterer J. A Probable Life-Saving Switch from Apixaban to Phenprocoumon. Heart Surg Forum. 2015 Oct 28;18(5):E186-7. doi: 10.1532/hsf.1268. PMID 26509341
- [Background] Caldeira D, Goncalves N, Pinto FJ, Costa J, Ferreira JJ. Risk of renal failure with the non-vitamin K antagonist oral anticoagulants: systematic review and meta-analysis. Pharmacoepidemiol Drug Saf. 2015 Jul;24(7):757-64. doi: 10.1002/pds.3791. Epub 2015 May 23. PMID 26009864
- [Background] ROCKET AF Study Investigators. Rivaroxaban-once daily, oral, direct factor Xa inhibition compared with vitamin K antagonism for prevention of stroke and Embolism Trial in Atrial Fibrillation: rationale and design of the ROCKET AF study. Am Heart J. 2010 Mar;159(3):340-347.e1. doi: 10.1016/j.ahj.2009.11.025. PMID 20211293
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Bohm M, Ezekowitz MD, Connolly SJ, Eikelboom JW, Hohnloser SH, Reilly PA, Schumacher H, Brueckmann M, Schirmer SH, Kratz MT, Yusuf S, Diener HC, Hijazi Z, Wallentin L. Changes in Renal Function in Patients With Atrial Fibrillation: An Analysis From the RE-LY Trial. J Am Coll Cardiol. 2015 Jun 16;65(23):2481-93. doi: 10.1016/j.jacc.2015.03.577. PMID 26065986
- [Background] Eriksson BI, Borris LC, Friedman RJ, Haas S, Huisman MV, Kakkar AK, Bandel TJ, Beckmann H, Muehlhofer E, Misselwitz F, Geerts W; RECORD1 Study Group. Rivaroxaban versus enoxaparin for thromboprophylaxis after hip arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2765-75. doi: 10.1056/NEJMoa0800374. PMID 18579811

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: 8 patients were enrolled in the study. Baseline creatinine and urinalysis was obtained.
Period: Overall Study
Arm/Group | Participants
Started | 8
Completed | 0
Not Completed | 8
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Anticoagulant-related Nephropathy in the Cohort
Description: Primary endpoint - Incidence of ARN is the primary outcome of this study and this is based on a documentation of AKI (defined as an increase in baseline serum creatinine ≥ 0.3 mg/dL), in the absence of any other obvious etiology for the AKI identified after a standard clinical evaluation and work up by the patient's primary care physician, cardiologist or nephrologist. This incidence will be expressed as a percentage.
Time Frame: 6 months
Measure: Number; unit: Percentage of participants
Arm/Group | Participants
Number analyzed (Participants) | 8
Percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: This is a prospective observational study. The study did not administer any treatment/interventions for patients. The patients kidney function and urinalysis were observed while they were on anticoagulation.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
The reference section is accurate and is not meant to be related to our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-07-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT02900170/Prot_000.pdf